CLINICAL TRIAL: NCT00303628
Title: Intergroup Randomized Phase III Study of Postoperative Oxaliplatin, 5-Fluorouracil and Leucovorin vs Oxaliplatin, 5-Fluorouracil, Leucovorin and Bevacizumab for Patients With Stage II or III Rectal Cancer Receiving Pre-operative Chemoradiation
Brief Title: Postoperative Chemotherapy With or Without Bevacizumab for Patients With Stage II or III Rectal Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was terminated before reaching its accrual goal due to slow accrual.
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E5204; NCI-2009-00563 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000467561 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); E5204 (Other: ECOG-ACRIN Cancer Research Group); U10CA021115 (NIH)
Record Dates: First submitted 2006-03-15; First posted 2006-03-17 (Estimated); Results first posted 2016-02-26 (Estimated); Last update posted 2023-07-06 (Actual); Status verified 2023-06

CONDITIONS: Adenocarcinoma of the Rectum; Stage II Rectal Cancer; Stage III Rectal Cancer
Keywords: Rectal cancer; Bevacizumab
MeSH Terms: conditions — Rectal Neoplasms | interventions — Oxaliplatin; Fluorouracil; Leucovorin; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (Active Comparator): Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV on day 1 followed by fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment repeats every 2 weeks for up to 12 courses.
  Interventions: Drug: oxaliplatin; Drug: fluorouracil; Drug: leucovorin calcium
- Arm II (Experimental): Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive oxaliplatin, leucovorin calcium, and fluorouracil as in arm I.
  Interventions: Drug: oxaliplatin; Drug: fluorouracil; Drug: leucovorin calcium; Drug: bevacizumab

INTERVENTIONS:
Drug: oxaliplatin — Given IV
  Other Names: 1-OHP; Dacotin; Dacplat; Eloxatin; L-OHP
Drug: fluorouracil — Given IV
  Other Names: 5-fluorouracil; 5-Fluracil; 5-FU
Drug: leucovorin calcium — Given IV
  Other Names: CF; CFR; LV
Drug: bevacizumab — Given IV
  Other Names: anti-VEGF humanized monoclonal antibody; anti-VEGF monoclonal antibody; Avastin; rhuMAb VEGF
  Arms: Arm II

SUMMARY:
Drugs used in chemotherapy, such as oxaliplatin, leucovorin, and fluorouracil, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Monoclonal antibodies, such as bevacizumab, can block tumor growth in different ways. Some block the ability of tumor cells to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Bevacizumab may also stop the growth of tumor cells by blocking blood flow to the tumor. Giving more than one drug (combination chemotherapy) together with bevacizumab after surgery may kill any tumor cells that remain after surgery. It is not yet known whether oxaliplatin, leucovorin, and fluorouracil is more effective with or without bevacizumab in treating rectal cancer. This randomized phase III trial is studying combination chemotherapy to see how well it works with or without bevacizumab in treating patients who have had surgery for stage II or stage III rectal cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Compare the overall survival of patients who have undergone prior surgery and neoadjuvant chemoradiotherapy for clinical stage II or III rectal cancer treated with adjuvant oxaliplatin, leucovorin calcium, fluorouracil with vs without bevacizumab.

SECONDARY OBJECTIVES:

I. Evaluate tolerance of treatment, patterns of failure, and disease-free survival in patients treated with these regimens

EXPLORATORY OBJECTIVES:

I. Assess long-term rectal function using the Patient Bowel Function/Uniscale questionnaire and the Functional Assessment of Cancer (FACT)-Diarrhea subscale in patients treated with these regimens.

II. Validate the FACT-Diarrhea subscale. III. Assess long-term symptoms of oxaliplatin-related neurotoxicity using the FACT/Gynecologic Oncology Group (GOG)-Neurotoxicity subscale in patients treated with these regimens.

IV. Correlate TS, DPD and TP expression (key targets for fluorouracil); retention of chromosome 18q alleles and microsatellite instability (MSI) with TGFβ1RII mutation (markers for fluorouracil efficacy); ERCC1, ERCC2, and XPF expression (participants in repair of adducts from oxaliplatin); and p53 gene mutation and possibly other molecular markers pertinent to vascular endothelial growth factor in tumor tissue specimens with treatment efficacy in these patients.

V. Correlate tumor molecular prognostic markers (chromosome 18q allelic loss and MSI) with survival in patients treated with this regimen.

OUTLINE:

This is a randomized study. Patients are stratified according to Eastern Cooperative Oncology Group (ECOG) performance status (0 vs 1), clinical staging (high risk [T3, N+, M0 or T4, any N, M0] vs low risk [T1-2, N+, M0 or T3, N0, M0]), prior pre-operative oxaliplatin (yes vs no), and prior radiotherapy dose (40-50 Gy vs > 50-55.8 Gy). Patients are randomized to 1 of 2 treatment arms in a 1:1 ratio.

ARM I: Patients receive oxaliplatin intravenously (IV) over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV on day 1 followed by fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment repeats every 2 weeks for up to 12 courses* in the absence of disease progression or unacceptable toxicity.

ARM II: Patients receive bevacizumab** IV over 30-90 minutes on day 1. Patients also receive oxaliplatin, leucovorin calcium, and fluorouracil as in arm I*.

[Note: *Patients who received prior neoadjuvant oxaliplatin including patients on protocol NSABP-R-04 receive up to 9 courses of treatment followed by leucovorin calcium IV and fluorouracil IV with (arm II) or without (arm I) bevacizumab for up to 3 courses.]

[Note: **Patients no longer receive bevacizumab as of 4/29/2009 when accrual was terminated due to slow accrual for the study)]

Patients complete 10-15 minute questionnaires about bowel function at randomization, end of treatment, 12 months post-treatment and then annually to 5 years post-treatment.

After completion of study treatment, patients are followed periodically for approximately 10 years.

PROJECTED ACCRUAL: 2100 patients

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed adenocarcinoma of the rectum meeting 1 of the following clinical (e.g., before neoadjuvant therapy) or pathologic staging criteria:

  * T3, N+, M0
  * T3, N0, M0
  * T4, N0, M0
  * Any T, N1-2, M0
* T4, N0-2, M0 disease must meet 1 of the following criteria:

  * Clinically fixed tumor on rectal examination with tumor adherent to the pelvic sidewall or sacrum
  * Hydronephrosis on Computed Tomography (CT) scan or Intravenous Pyelogram (IVP)
  * Ureteric or bladder invasion as documented by cystoscopy and cytology or biopsy
  * Invasion into prostate
  * Vaginal or uterine involvement
* Must have undergone complete tumor resection >= 28 days ago and able to begin treatment by day 56
* Must have undergone concurrent neoadjuvant chemoradiotherapy*

  * NOTE: *Neoadjuvant chemoradiotherapy received on protocol NSABP-R-04 allowed provided it met these criteria
* Must have undergone prior radiotherapy at 40-55.8 Gy** AND received 1 of the following chemotherapy regimens:

  * Continuous infusion of fluorouracil with or without oxaliplatin; fluorouracil and leucovorin calcium
  * Capecitabine with or without oxaliplatin; capecitabine with or without oxaliplatin OR a continuous infusion of fluorouracil with or without oxaliplatin received on protocol NSABP-R-04
  * NOTE: **Intensity-modulated radiotherapy allowed
* ECOG performance status 0-1
* Platelet count >= 100,000/mm^3
* Absolute granulocyte count >= 1,500/mm^3
* Bilirubin normal (unless chronic grade 1 bilirubin elevation due to Gilbert's disease or similar syndrome due to slow conjugation of bilirubin)
* Alkaline phosphatase (AP) < 2.5 times upper limit of normal (ULN) and aspartate aminotransferase (AST) < 1.5 times ULN
* Hepatitis B and C negative (for patients with AP > normal) unless previously vaccinated
* Serum creatinine =< 1.5 times ULN
* Urine protein:creatinine (UPC) ratio < 1.0 OR urine protein < 1 g on 24-hour urine collection
* International Normalized Ratio (INR) =< 1.5
* INR > 1.5 allowed provided patient is on full-dose anticoagulants AND meets all of the following criteria:

  * In-range INR (i.e., between 2 and 3) on a stable dose of warfarin or low molecular weight heparin
  * No active bleeding or pathological condition that is associated with a high risk of bleeding
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 3 months after study treatment
* No other previous or concurrent malignancy except nonmelanoma skin cancer, breast cancer in situ, carcinoma in situ of the cervix, or previously treated nonpelvic cancer that has been disease-free for > 5 years
* Patients with a history of breast cancer (without evidence of disease) who remain on hormonal therapy for > 5 years are eligible
* Patients with a history of hypertension must have blood pressure < 150/90 mm Hg AND be on a stable regimen of antihypertensive therapy
* No other prior chemotherapy or pelvic radiotherapy except as neoadjuvant treatment for current diagnosis of rectal cancer
* Concurrent participation on protocol NSABP-R-04 allowed

Exclusion Criteria:

* Pregnant or nursing
* Evidence of metastatic disease on the surgical/intraoperative examination
* Evidence of metastatic disease confirmed by CT scan, Magnetic resonance imaging (MRI), or ultrasound of the liver or chest CT scan or chest x-ray within the past 6 months
* Evidence of tumor outside of the pelvis, including liver metastases, peritoneal seeding, or metastatic inguinal lymphadenopathy
* Concurrent major surgery
* Active bleeding not related to the primary rectal tumor within the past 6 months
* Active inflammatory bowel disease or other serious medical illness which might limit the ability of the patient to receive protocol therapy
* Active gastroduodenal ulcer determined by endoscopy
* Serious or nonhealing wound, skin ulcer, or bone fracture
* Clinically significant peripheral sensory or motor neuropathy >= grade 2
* Nonmalignant systemic disease (e.g., cardiovascular, renal, or hepatic) that would preclude study treatment including, but not limited to, any of the following:

  * New York Heart Association class III or IV congestive heart failure
  * Concurrent symptomatic arrhythmia
* Transient ischemic attack or cerebrovascular accident
* Arterial thromboembolic event, unstable angina, or myocardial infarction within the past 12 months
* Significant peripheral vascular disease
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude study requirements
* Significant traumatic injury within the past 28 days
* Known allergy to platinum compounds
* Prior invasive procedure, including either of the following:

  * Major surgical procedure or open biopsy within the past 28 days
  * Core biopsy or other minor procedure, except placement of a vascular access device, within the past 7 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 355 (Actual)
Dates: Start 2006-05-11 (Actual); Primary Completion 2015-04 (Actual); Study Completion 2019-02-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Al Benson, Principal Investigator — Eastern Cooperative Oncology Group
Locations (617):
- United States (600):
  - Providence Hospital, Mobile, Alabama
  - Providence Alaska Medical Center, Anchorage, Alaska
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Saint Bernards Regional Medical Center, Jonesboro, Arkansas
  - Alta Bates Summit Medical Center-Herrick Campus, Berkeley, California
  - Mills - Peninsula Hospitals, Burlingame, California
  - East Bay Radiation Oncology Center, Castro Valley, California
  - Eden Hospital Medical Center, Castro Valley, California
  - Valley Medical Oncology Consultants-Castro Valley, Castro Valley, California
  - Kaiser Permanente, Fremont, Fremont, California
  - Valley Medical Oncology Consultants-Fremont, Fremont, California
  - Cancer Care Associates of Fresno Medical Group Inc, Fresno, California
  - Saint Jude Medical Center, Fullerton, California
  - Glendale Memorial Hospital and Health Center, Glendale, California
  - Marin General Hospital, Greenbrae, California
  - Kaiser Permanente, Hayward, Hayward, California
  - Saint Rose Hospital, Hayward, California
  - University of Southern California/Norris Cancer Center, Los Angeles, California
  - Contra Costa Regional Medical Center, Martinez, California
  - Fremont - Rideout Cancer Center, Marysville, California
  - Community Hospital of Monterey Peninsula, Monterey, California
  - El Camino Hospital, Mountain View, California
  - Palo Alto Medical Foundation-Camino Division, Mountain View, California
  - Sutter Cancer Research Consortium, Novato, California
  - Highland General Hospital, Oakland, California
  - Alta Bates Summit Medical Center - Summit Campus, Oakland, California
  - Bay Area Breast Surgeons Inc, Oakland, California
  - Bay Area Tumor Institute CCOP, Oakland, California
  - Larry G Strieff MD Medical Corporation, Oakland, California
  - Tom K Lee Inc, Oakland, California
  - Kaiser Permanente-Oakland, Oakland, California
  - Desert Regional Medical Center, Palm Springs, California
  - Palo Alto Medical Foundation Heath Care, Palo Alto, California
  - Valley Care Health System - Pleasanton, Pleasanton, California
  - Valley Medical Oncology Consultants, Pleasanton, California
  - Kaiser Permanente-Redwood City, Redwood City, California
  - Kaiser Permanente-Richmond, Richmond, California
  - Kaiser Permanente-Roseville, Roseville, California
  - University of California at Davis Cancer Center, Sacramento, California
  - Kaiser Permanente-South Sacramento, Sacramento, California
  - Kaiser Permanente - Sacramento, Sacramento, California
  - Salinas Valley Memorial, Salinas, California
  - University of California At San Diego, San Diego, California
  - Kaiser Permanente, San Diego, California
  - Kaiser Permanente-San Francisco, San Francisco, California
  - California Pacific Medical Center, San Francisco, California
  - Kaiser Permanente-Santa Teresa-San Jose, San Jose, California
  - Doctors Medical Center- JC Robinson Regional Cancer Center, San Pablo, California
  - Kaiser Permanente-San Rafael, San Rafael, California
  - Kaiser Permanente Medical Center - Santa Clara, Santa Clara, California
  - Kaiser Permanente-Santa Rosa, Santa Rosa, California
  - Kaiser Permanente-South San Francisco, South San Francisco, California
  - Kaiser Permanente-Stockton, Stockton, California
  - Tahoe Forest Cancer Center, Truckee, California
  - Kaiser Permanente-Vallejo, Vallejo, California
  - Sutter Solano Medical Center, Vallejo, California
  - Kaiser Permanente-Walnut Creek, Walnut Creek, California
  - The Medical Center of Aurora, Aurora, Colorado
  - Boulder Community Hospital, Boulder, Colorado
  - Penrose-Saint Francis Healthcare, Colorado Springs, Colorado
  - Memorial Hospital Colorado Springs, Colorado Springs, Colorado
  - Porter Adventist Hospital, Denver, Colorado
  - Exempla Saint Joseph Hospital, Denver, Colorado
  - Presbyterian - Saint Lukes Medical Center - Health One, Denver, Colorado
  - Rose Medical Center, Denver, Colorado
  - Colorado Cancer Research Program CCOP, Denver, Colorado
  - Swedish Medical Center, Englewood, Colorado
  - Front Range Cancer Specialists, Fort Collins, Colorado
  - Saint Mary's Hospital and Regional Medical Center, Grand Junction, Colorado
  - North Colorado Medical Center, Greeley, Colorado
  - Saint Anthony Hospital, Lakewood, Colorado
  - Sky Ridge Medical Center, Lone Tree, Colorado
  - Longmont United Hospital, Longmont, Colorado
  - McKee Medical Center, Loveland, Colorado
  - Saint Mary Corwin Medical Center, Pueblo, Colorado
  - North Suburban Medical Center, Thornton, Colorado
  - Exempla Lutheran Medical Center, Wheat Ridge, Colorado
  - Eastern Connecticut Hematology and Oncology Associates, Norwich, Connecticut
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Washington Hospital Center, Washington D.C., District of Columbia
  - Lombardi Comprehensive Cancer Center at Georgetown University, Washington D.C., District of Columbia
  - Holy Cross Hospital, Fort Lauderdale, Florida
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Jupiter Medical Center, Jupiter, Florida
  - The Watson Clinic, Lakeland, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - Mount Sinai Medical Center CCOP, Miami Beach, Florida
  - Cancer Specialists of North Florida-Orange Park, Orange Park, Florida
  - University Cancer and Blood Center LLC, Athens, Georgia
  - Piedmont Hospital, Atlanta, Georgia
  - Atlanta Regional CCOP, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Saint Joseph's Hospital of Atlanta, Atlanta, Georgia
  - Georgia Regents University, Augusta, Georgia
  - Well Star Cobb Hospital, Austell, Georgia
  - Atlanta VA Medical Center, Decatur, Georgia
  - Dekalb Medical Center, Decatur, Georgia
  - Gwinnett Medical Center, Lawrenceville, Georgia
  - Medical Center of Central Georgia, Macon, Georgia
  - Wellstar Kennestone Hospital, Marietta, Georgia
  - Southern Regional Medical Center, Riverdale, Georgia
  - Harbin Clinic Medical Oncology and Clinical Research, Rome, Georgia
  - Memorial Health University Medical Center, Savannah, Georgia
  - Oncare Hawaii Inc-POB II, Honolulu, Hawaii
  - Queen's Medical Center, Honolulu, Hawaii
  - Straub Clinic and Hospital, Honolulu, Hawaii
  - University of Hawaii, Honolulu, Hawaii
  - Oncare Hawaii Inc-Kuakini, Honolulu, Hawaii
  - The Cancer Center of Hawaii-Liliha, Honolulu, Hawaii
  - Kapiolani Medical Center for Women and Children, Honolulu, Hawaii
  - Tripler Army Medical Center, Honolulu, Hawaii
  - Maui Memorial Medical Center, Wailuku, Hawaii
  - Pacific Cancer Institute of Maui, Wailuku, Hawaii
  - Pali Momi Medical Center, ‘Aiea, Hawaii
  - Saint Alphonsus Regional Medical Center, Boise, Idaho
  - Saint Luke's Mountain States Tumor Institute, Boise, Idaho
  - Hematology Oncology Associates of Eastern Idaho, Idaho Falls, Idaho
  - Portneuf Medical Center, Pocatello, Idaho
  - Saint Anthony's Health, Alton, Illinois
  - Rush - Copley Medical Center, Aurora, Illinois
  - Saint Joseph Medical Center, Bloomington, Illinois
  - Graham Hospital Association, Canton, Illinois
  - Memorial Hospital, Carthage, Illinois
  - Mount Sinai Hospital Medical Center, Chicago, Illinois
  - Hematology and Oncology Associates, Chicago, Illinois
  - Northwestern University, Chicago, Illinois
  - John H Stroger Jr Hospital of Cook County, Chicago, Illinois
  - Jesse Brown Veterans Affairs Medical Center, Chicago, Illinois
  - Rush University Medical Center, Chicago, Illinois
  - Mercy Hospital and Medical Center, Chicago, Illinois
  - Swedish Covenant Hospital, Chicago, Illinois
  - Resurrection Healthcare, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Decatur Memorial Hospital, Decatur, Illinois
  - Good Samaritan Hospital, Downers Grove, Illinois
  - Elmhurst Memorial Hospital, Elmhurst, Illinois
  - Eureka Hospital, Eureka, Illinois
  - NorthShore University HealthSystem-Evanston Hospital, Evanston, Illinois
  - Saint Francis Hospital, Evanston, Illinois
  - Galesburg Cottage Hospital, Galesburg, Illinois
  - Illinois CancerCare Galesburg, Galesburg, Illinois
  - Western Illinois Cancer Treatment Center, Galesburg, Illinois
  - Mason District Hospital, Havana, Illinois
  - Hinsdale Hematology Oncology Associates Incorporated, Hinsdale, Illinois
  - Hopedale Medical Complex - Hospital, Hopedale, Illinois
  - Midwest Center for Hematology Oncology, Joliet, Illinois
  - Joliet Oncology-Hematology Associates Limited, Joliet, Illinois
  - Kewanee Hospital, Kewanee, Illinois
  - North Shore Hematology Oncology, Libertyville, Illinois
  - Mcdonough District Hospital, Macomb, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Garneau, Stewart C MD (UIA Investigator), Moline, Illinois
  - Porubcin, Michael MD (UIA Investigator), Moline, Illinois
  - Sharis, Christine M MD (UIA Investigator), Moline, Illinois
  - Stoffel, Thomas J MD (UIA Investigator), Moline, Illinois
  - Vigliotti, Antonio, P.G. M.D. (UIA Investigator), Moline, Illinois
  - Good Samaritan Regional Health Center, Mount Vernon, Illinois
  - Edward Hospital/Cancer Center, Naperville, Illinois
  - Illinois Cancer Specialists-Niles, Niles, Illinois
  - Bromenn Regional Medical Center, Normal, Illinois
  - Community Cancer Center Foundation, Normal, Illinois
  - Illinois CancerCare-Ottawa Clinic, Ottawa, Illinois
  - Ottawa Regional Hospital and Healthcare Center, Ottawa, Illinois
  - Pekin Cancer Treatment Center, Pekin, Illinois
  - Pekin Hospital, Pekin, Illinois
  - Methodist Medical Center of Illinois, Peoria, Illinois
  - Proctor Hospital, Peoria, Illinois
  - OSF Saint Francis Medical Center Radiation Oncology Service at the Central Illinois Comprehensive CC, Peoria, Illinois
  - Illinois CancerCare-Peoria, Peoria, Illinois
  - Illinois Oncology Research Association CCOP, Peoria, Illinois
  - OSF Saint Francis Medical Center, Peoria, Illinois
  - Illinois Valley Hospital, Peru, Illinois
  - Valley Radiation Oncology, Peru, Illinois
  - Perry Memorial Hospital, Princeton, Illinois
  - Swedish American Hospital, Rockford, Illinois
  - Edward H Kaplan MD and Associates, Skokie, Illinois
  - Hematology Oncology Associates of Illinois - Skokie, Skokie, Illinois
  - Midwest Cancer Research Group Incorporated, Skokie, Illinois
  - Saint Margaret's Hospital, Spring Valley, Illinois
  - Memorial Medical Center, Springfield, Illinois
  - Carle Cancer Center, Urbana, Illinois
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Saint Francis Hospital and Health Centers, Beech Grove, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Fort Wayne Medical Oncology and Hematology Inc-Parkview, Fort Wayne, Indiana
  - Saint Vincent Hospital and Health Services, Indianapolis, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Franciscan Saint Anthony Health-Michigan City, Michigan City, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - IU Health Ball Memorial Hospital, Muncie, Indiana
  - Oncology Hematology Associates of Southwest Indiana, Newburgh, Indiana
  - Reid Hospital and Health Care Services, Richmond, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - McFarland Clinic PC-William R Bliss Cancer Center, Ames, Iowa
  - Constantinou, Costas L MD (UIA Investigator), Bettendorf, Iowa
  - Cedar Rapids Oncology Association, Cedar Rapids, Iowa
  - Oncology Associates at Mercy Medical Center, Cedar Rapids, Iowa
  - Medical Oncology and Hematology Associates-West Des Moines, Clive, Iowa
  - Genesis Medical Center - East Campus, Davenport, Iowa
  - Genesis Medical Center - West Campus, Davenport, Iowa
  - Mercy Capitol, Des Moines, Iowa
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Iowa Oncology Research Association CCOP, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Des Moines, Des Moines, Iowa
  - Medical Oncology and Hematology Associates-Laurel, Des Moines, Iowa
  - Mercy Medical Center - Des Moines, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Mercy Medical Center - North Iowa, Mason City, Iowa
  - Siouxland Regional Cancer Center, Sioux City, Iowa
  - Siouxland Hematology Oncology Associates, Sioux City, Iowa
  - Mercy Medical Center-Sioux City, Sioux City, Iowa
  - Saint Luke's Regional Medical Center, Sioux City, Iowa
  - Cedar Valley Medical Specialists, Waterloo, Iowa
  - Covenant Medical Center, Waterloo, Iowa
  - Hospital District Sixth of Harper County, Anthony, Kansas
  - Cancer Center of Kansas - Chanute, Chanute, Kansas
  - Cancer Center of Kansas - Dodge City, Dodge City, Kansas
  - Cancer Center of Kansas - El Dorado, El Dorado, Kansas
  - Cancer Center of Kansas - Fort Scott, Fort Scott, Kansas
  - Cancer Center of Kansas-Independence, Independence, Kansas
  - University of Kansas Medical Center, Kansas City, Kansas
  - Cancer Center of Kansas-Kingman, Kingman, Kansas
  - Lawrence Memorial Hospital, Lawrence, Kansas
  - Cancer Center of Kansas - Newton, Newton, Kansas
  - Olathe Cancer Center, Olathe, Kansas
  - Cancer Center of Kansas - Parsons, Parsons, Kansas
  - Cancer Center of Kansas - Pratt, Pratt, Kansas
  - Cancer Center of Kansas - Salina, Salina, Kansas
  - Stormont-Vail Regional Health Center, Topeka, Kansas
  - Cancer Center of Kansas - Wellington, Wellington, Kansas
  - Associates In Womens Health, Wichita, Kansas
  - Cancer Center of Kansas-Wichita Medical Arts Tower, Wichita, Kansas
  - Cancer Center of Kansas - Main Office, Wichita, Kansas
  - Via Christi Regional Medical Center, Wichita, Kansas
  - Wichita CCOP, Wichita, Kansas
  - Cancer Center of Kansas - Winfield, Winfield, Kansas
  - The James Graham Brown Cancer Center at University of Louisville, Louisville, Kentucky
  - Eastern Maine Medical Center, Bangor, Maine
  - Saint Mary's Regional Medical Center, Lewiston, Maine
  - Maine Medical Center- Scarborough Campus, Scarborough, Maine
  - Franklin Square Hospital Center, Baltimore, Maryland
  - Memorial Hospital at Easton - Shore Regional Cancer Center, Easton, Maryland
  - Union Hospital of Cecil County, Elkton, Maryland
  - Eastern Cooperative Oncology Group, Boston, Massachusetts
  - Caritas Saint Elizabeth's Medical Center, Brighton, Massachusetts
  - Lahey Hospital and Medical Center, Burlington, Massachusetts
  - Simonds-Sinon Regional Cancer Center, Fitchburg, Massachusetts
  - Berkshire Hematology Oncology PC, Pittsfield, Massachusetts
  - University of Massachusetts Medical School, Worcester, Massachusetts
  - Bixby Medical Center, Adrian, Michigan
  - Hickman Cancer Center, Adrian, Michigan
  - Saint Joseph Mercy Hospital, Ann Arbor, Michigan
  - Michigan Cancer Research Consortium Community Clinical Oncology Program, Ann Arbor, Michigan
  - Bronson Battle Creek, Battle Creek, Michigan
  - Spectrum Health Big Rapids Hospital, Big Rapids, Michigan
  - Oakwood Hospital, Dearborn, Michigan
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - Saint John Hospital and Medical Center, Detroit, Michigan
  - Green Bay Oncology - Escanaba, Escanaba, Michigan
  - Hurley Medical Center, Flint, Michigan
  - Genesys Regional Medical Center-West Flint Campus, Flint, Michigan
  - Grand Rapids Clinical Oncology Program, Grand Rapids, Michigan
  - Mercy Health Saint Mary's, Grand Rapids, Michigan
  - Spectrum Health at Butterworth Campus, Grand Rapids, Michigan
  - Holland Community Hospital, Holland, Michigan
  - Green Bay Oncology - Iron Mountain, Iron Mountain, Michigan
  - Allegiance Health, Jackson, Michigan
  - Sparrow Hospital, Lansing, Michigan
  - Saint Mary Mercy Hospital, Livonia, Michigan
  - Marquette General Hospital, Marquette, Michigan
  - Community Cancer Center of Monroe, Monroe, Michigan
  - Mercy Memorial Hospital, Monroe, Michigan
  - Mercy Health Partners-Hackley Campus, Muskegon, Michigan
  - Mercy Health Mercy Campus, Muskegon, Michigan
  - Saint Joseph Mercy Oakland, Pontiac, Michigan
  - Saint Joseph Mercy Port Huron, Port Huron, Michigan
  - William Beaumont Hospital-Royal Oak, Royal Oak, Michigan
  - Saint Mary's of Michigan, Saginaw, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Munson Medical Center, Traverse City, Michigan
  - Saint John Macomb-Oakland Hospital, Warren, Michigan
  - Metro Health Hospital, Wyoming, Michigan
  - Sanford Clinic North-Bemidgi, Bemidji, Minnesota
  - Fairview Ridges Hospital, Burnsville, Minnesota
  - Mercy Hospital, Coon Rapids, Minnesota
  - Essentia Health Duluth Clinic CCOP, Duluth, Minnesota
  - Essentia Health Saint Mary's Medical Center, Duluth, Minnesota
  - Miller-Dwan Hospital, Duluth, Minnesota
  - Fairview-Southdale Hospital, Edina, Minnesota
  - Unity Hospital, Fridley, Minnesota
  - Hutchinson Area Health Care, Hutchinson, Minnesota
  - Meeker County Memorial Hospital, Litchfield, Minnesota
  - Mayo Clinic Health Systems-Mankato, Mankato, Minnesota
  - Minnesota Oncology Hematology PA-Maplewood, Maplewood, Minnesota
  - Saint John's Hospital - Healtheast, Maplewood, Minnesota
  - Abbott-Northwestern Hospital, Minneapolis, Minnesota
  - Virginia Piper Cancer Institute, Minneapolis, Minnesota
  - Hennepin County Medical Center, Minneapolis, Minnesota
  - Minneapolis Veterans Medical Center, Minneapolis, Minnesota
  - North Memorial Medical Health Center, Robbinsdale, Minnesota
  - Mayo Clinic, Rochester, Minnesota
  - Metro-Minnesota CCOP, Saint Louis Park, Minnesota
  - Park Nicollet Clinic - Saint Louis Park, Saint Louis Park, Minnesota
  - Regions Hospital, Saint Paul, Minnesota
  - Saint Joseph's Hospital - Healtheast, Saint Paul, Minnesota
  - United Hospital, Saint Paul, Minnesota
  - Saint Francis Regional Medical Center, Shakopee, Minnesota
  - Ridgeview Medical Center, Waconia, Minnesota
  - Rice Memorial Hospital, Willmar, Minnesota
  - Minnesota Oncology and Hematology PA-Woodbury, Woodbury, Minnesota
  - Woodwinds Health Campus, Woodbury, Minnesota
  - Southeast Missouri Hospital, Cape Girardeau, Missouri
  - Saint Francis Medical Center, Cape Girardeau, Missouri
  - Freeman Health System, Joplin, Missouri
  - Mercy Hospital-Joplin, Joplin, Missouri
  - Mercy Hospital Springfield, Springfield, Missouri
  - CoxHealth South Hospital, Springfield, Missouri
  - Saint Louis Cancer and Breast Institute-South City, St Louis, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Missouri Baptist Medical Center, St Louis, Missouri
  - Center for Cancer Care and Research, St Louis, Missouri
  - Saint John's Mercy Medical Center, St Louis, Missouri
  - Saint Louis-Cape Girardeau CCOP, St Louis, Missouri
  - Montana Cancer Consortium CCOP, Billings, Montana
  - Northern Rockies Radiation Oncology Center, Billings, Montana
  - Saint Vincent Healthcare, Billings, Montana
  - Hematology-Oncology Centers of the Northern Rockies PC, Billings, Montana
  - Billings Clinic, Billings, Montana
  - Deaconess Medical Center, Billings, Montana
  - Bozeman Deaconess Cancer Center, Bozeman, Montana
  - Bozeman Deaconess Hospital, Bozeman, Montana
  - Saint James Community Hospital and Cancer Treatment Center, Butte, Montana
  - Benefis Healthcare- Sletten Cancer Institute, Great Falls, Montana
  - Berdeaux, Donald MD (UIA Investigator), Great Falls, Montana
  - Great Falls Clinic, Great Falls, Montana
  - Northern Montana Hospital, Havre, Montana
  - Saint Peter's Community Hospital, Helena, Montana
  - Glacier Oncology PLLC, Kalispell, Montana
  - Kalispell Medical Oncology, Kalispell, Montana
  - Kalispell Regional Medical Center, Kalispell, Montana
  - Community Medical Hospital, Missoula, Montana
  - Montana Cancer Specialists, Missoula, Montana
  - Saint Patrick Hospital - Community Hospital, Missoula, Montana
  - Guardian Oncology and Center for Wellness, Missoula, Montana
  - Nebraska Cancer Research Center, Lincoln, Nebraska
  - Missouri Valley Cancer Consortium CCOP, Omaha, Nebraska
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - Alegent Health Immanuel Medical Center, Omaha, Nebraska
  - Alegent Health Bergan Mercy Medical Center, Omaha, Nebraska
  - Creighton University Medical Center, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - University Medical Center of Southern Nevada, Las Vegas, Nevada
  - Nevada Cancer Research Foundation CCOP, Las Vegas, Nevada
  - Exeter Hospital, Exeter, New Hampshire
  - Cheshire Medical Center-Dartmouth-Hitchcock Keene, Keene, New Hampshire
  - Elliot Hospital, Manchester, New Hampshire
  - Ocean Medical Center, Brick, New Jersey
  - Cooper Hospital University Medical Center, Camden, New Jersey
  - Cancer Institute of New Jersey At Hamilton, Hamilton, New Jersey
  - Monmouth Medical Center, Long Branch, New Jersey
  - Mountainside Hospital, Montclair, New Jersey
  - Morristown Memorial Hospital, Morristown, New Jersey
  - Fox Chase Cancer Center at Virtua Memorial Hospital of Burlington County, Mount Holly, New Jersey
  - Rutgers Cancer Institute of New Jersey, New Brunswick, New Jersey
  - Newark Beth Israel Medical Center, Newark, New Jersey
  - Valley Hospital, Ridgewood, New Jersey
  - Sparta Cancer Treatment Center, Sparta, New Jersey
  - Overlook Hospital, Summit, New Jersey
  - Virtua West Jersey Hospital Voorhees, Voorhees Township, New Jersey
  - Hematology Oncology Associates, Albuquerque, New Mexico
  - University of New Mexico Cancer Center, Albuquerque, New Mexico
  - Presbyterian Kaseman Hospital, Albuquerque, New Mexico
  - New Mexico Cancer Care Associates, Santa Fe, New Mexico
  - Kings County Hospital, Brooklyn, New York
  - State University of New York Downstate Medical Center, Brooklyn, New York
  - University Hospital of Brooklyn, Brooklyn, New York
  - Veterans Affairs Western New York Health Care System-Buffalo, Buffalo, New York
  - Roswell Park Cancer Institute, Buffalo, New York
  - Hematology Oncology Associates of Central New York PC-East Syracuse, East Syracuse, New York
  - Glens Falls Hospital, Glens Falls, New York
  - Orange Regional Medical Center, Middletown, New York
  - New York University Langone Medical Center, New York, New York
  - Columbia University Medical Center, New York, New York
  - Weill Medical College of Cornell University, New York, New York
  - Highland Hospital, Rochester, New York
  - Interlakes Foundation Inc-Rochester, Rochester, New York
  - University of Rochester, Rochester, New York
  - State University of New York Upstate Medical University, Syracuse, New York
  - Community General Hospital, Syracuse, New York
  - Albert Einstein College of Medicine, The Bronx, New York
  - Montefiore Medical Center, The Bronx, New York
  - Mission Hospital-Memorial Campus, Asheville, North Carolina
  - Cone Health Alamance Regional Medical Center, Burlington, North Carolina
  - Carolinas Medical Center, Charlotte, North Carolina
  - Carolinas Medical Center - Northeast, Concord, North Carolina
  - Wayne Memorial Hospital, Goldsboro, North Carolina
  - Wayne Radiation Oncology, Goldsboro, North Carolina
  - Rutherford Hospital, Rutherfordton, North Carolina
  - Wilson Medical Center, Wilson, North Carolina
  - Bismarck Cancer Center, Bismarck, North Dakota
  - Mid Dakota Clinic, Bismarck, North Dakota
  - Saint Alexius Medical Center, Bismarck, North Dakota
  - Sanford Bismarck Medical Center, Bismarck, North Dakota
  - Sanford Clinic North-Fargo, Fargo, North Dakota
  - Sanford Medical Center-Fargo, Fargo, North Dakota
  - Altru Cancer Center, Grand Forks, North Dakota
  - Mary Rutan Hospital, Bellefontaine, Ohio
  - Toledo Clinic Cancer Centers-Bowling Green, Bowling Green, Ohio
  - Mercy Medical Center, Canton, Ohio
  - Aultman Health Foundation, Canton, Ohio
  - Adena Regional Medical Center, Chillicothe, Ohio
  - The Christ Hospital, Cincinnati, Ohio
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - MetroHealth Medical Center, Cleveland, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - North Coast Cancer Care-Clyde, Clyde, Ohio
  - Arthur G. James Cancer Hospital and Solove Research Institute at Ohio State University Medical Center, Columbus, Ohio
  - Riverside Methodist Hospital, Columbus, Ohio
  - Columbus CCOP, Columbus, Ohio
  - Grant Medical Center, Columbus, Ohio
  - Mount Carmel Health Center West, Columbus, Ohio
  - Doctors Hospital, Columbus, Ohio
  - Grandview Hospital, Dayton, Ohio
  - Good Samaritan Hospital - Dayton, Dayton, Ohio
  - Miami Valley Hospital, Dayton, Ohio
  - Samaritan North Health Center, Dayton, Ohio
  - Dayton CCOP, Dayton, Ohio
  - Veteran Affairs Medical Center, Dayton, Ohio
  - Grady Memorial Hospital, Delaware, Ohio
  - Hematology Oncology Center Incorporated, Elyria, Ohio
  - Blanchard Valley Hospital, Findlay, Ohio
  - Atrium Medical Center-Middletown Regional Hospital, Franklin, Ohio
  - Fremont Memorial Hospital, Fremont, Ohio
  - Wayne Hospital, Greenville, Ohio
  - Cleveland Clinic Cancer Center Independence, Independence, Ohio
  - Cole, Sharon, K. M.D. (UIA Investigator), Kenton, Ohio
  - Kettering Medical Center, Kettering, Ohio
  - Fairfield Medical Center, Lancaster, Ohio
  - Lima Memorial Hospital, Lima, Ohio
  - Marietta Memorial Hospital, Marietta, Ohio
  - Saint Luke's Hospital, Maumee, Ohio
  - Toledo Clinic Cancer Centers-Maumee, Maumee, Ohio
  - Toledo Radiation Oncology at Northwest Ohio Onocolgy Center, Maumee, Ohio
  - Licking Memorial Hospital, Newark, Ohio
  - Saint Charles Hospital, Oregon, Ohio
  - Toledo Clinic Cancer Centers-Oregon, Oregon, Ohio
  - Firelands Regional Medical Center, Sandusky, Ohio
  - North Coast Cancer Care, Sandusky, Ohio
  - Springfield Regional Medical Center, Springfield, Ohio
  - Flower Hospital, Sylvania, Ohio
  - Mercy Hospital of Tiffin, Tiffin, Ohio
  - The Toledo Hospital/Toledo Children's Hospital, Toledo, Ohio
  - Saint Vincent Mercy Medical Center, Toledo, Ohio
  - University of Toledo, Toledo, Ohio
  - Toledo Community Hospital Oncology Program CCOP, Toledo, Ohio
  - Mercy Saint Anne Hospital, Toledo, Ohio
  - Stark, Michael, Edward. M.D. (UIA Investigator), Toledo, Ohio
  - Toledo Clinic Cancer Centers-Toledo, Toledo, Ohio
  - Upper Valley Medical Center, Troy, Ohio
  - Fulton County Health Center, Wauseon, Ohio
  - Saint Ann's Hospital, Westerville, Ohio
  - Clinton Memorial Hospital, Wilmington, Ohio
  - Cleveland Clinic Wooster Specialty Center, Wooster, Ohio
  - Greene Memorial Hospital, Xenia, Ohio
  - Genesis HealthCare System, Zanesville, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Cancer Care Associates, Oklahoma City, Oklahoma
  - Natalie Warren Bryant Cancer Center at Saint Francis, Tulsa, Oklahoma
  - Saint Charles Medical Center-Bend, Bend, Oregon
  - Providence Milwaukie Hospital, Milwaukie, Oregon
  - Providence Portland Medical Center, Portland, Oregon
  - Western Oncology Research Consortium, Portland, Oregon
  - Adventist Medical Center, Portland, Oregon
  - Providence Saint Vincent Medical Center, Portland, Oregon
  - Kaiser Permanente, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - Saint Luke's University Hospital-Bethlehem Campus, Bethlehem, Pennsylvania
  - Bryn Mawr Hospital, Bryn Mawr, Pennsylvania
  - Geisinger Medical Center, Danville, Pennsylvania
  - Armstrong Center for Medicine and Health, Kittanning, Pennsylvania
  - Riddle Hospital, Media, Pennsylvania
  - Paoli Memorial Hospital, Paoli, Pennsylvania
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Albert Einstein Medical Center, Philadelphia, Pennsylvania
  - Allegheny Cancer Center at Allegheny General Hospital, Pittsburgh, Pennsylvania
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - Pottstown Memorial Medical Center, Pottstown, Pennsylvania
  - Mercy Hospital, Scranton, Pennsylvania
  - Hematology and Oncology Associates of North East Pennsylvania, Scranton, Pennsylvania
  - Scranton Hematology Oncology, Scranton, Pennsylvania
  - Geisinger Medical Group, State College, Pennsylvania
  - Reading Hospital, West Reading, Pennsylvania
  - Geisinger Wyoming Valley, Wilkes-Barre, Pennsylvania
  - Lankenau Hospital, Wynnewood, Pennsylvania
  - Mainline Health CCOP, Wynnewood, Pennsylvania
  - WellSpan Health-York Hospital, York, Pennsylvania
  - Hematology and Oncology Associates of Rhode Island Inc, Cranston, Rhode Island
  - Kent County Hospital, Warwick, Rhode Island
  - AnMed Health Hospital, Anderson, South Carolina
  - Roper Hospital, Charleston, South Carolina
  - McLeod Regional Medical Center, Florence, South Carolina
  - Greenville Health System Cancer Institute/Greenville CCOP, Greenville, South Carolina
  - Spartanburg Regional Medical Center, Spartanburg, South Carolina
  - Upstate Carolina CCOP, Spartanburg, South Carolina
  - Sanford Cancer Center-Oncology Clinic, Sioux Falls, South Dakota
  - Medical X-Ray Center, Sioux Falls, South Dakota
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Wellmont Holston Valley Hospital and Medical Center, Kingsport, Tennessee
  - Thompson Cancer Survival Center, Knoxville, Tennessee
  - University of Tennessee - Memphis, Memphis, Tennessee
  - Nashville Oncology Associates PC, Nashville, Tennessee
  - Tennessee Oncology PLLC- Centennial Medical Center, Nashville, Tennessee
  - Meharry Medical College, Nashville, Tennessee
  - Vanderbilt-Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - Zale Lipshy University Hospital, Dallas, Texas
  - Saint Paul Hospital, Dallas, Texas
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Tech University Health Sciences Center, Lubbock, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - American Fork Hospital, American Fork, Utah
  - Sandra L Maxwell Cancer Center, Cedar City, Utah
  - Logan Regional Hospital, Logan, Utah
  - Cottonwood Hospital Medical Center, Murray, Utah
  - Intermountain Medical Center, Murray, Utah
  - McKay-Dee Hospital Center, Ogden, Utah
  - Utah Valley Regional Medical Center, Provo, Utah
  - Intermountain Health Care, Salt Lake City, Utah
  - Utah Cancer Specialists-Salt Lake City, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah
  - LDS Hospital, Salt Lake City, Utah
  - Dixie Medical Center Regional Cancer Center, St. George, Utah
  - University of Vermont, Burlington, Vermont
  - Martha Jefferson Hospital, Charlottesville, Virginia
  - University of Virginia, Charlottesville, Virginia
  - Fredericksburg Oncology Inc, Fredericksburg, Virginia
  - Virginia Oncology Associates-Hampton, Hampton, Virginia
  - Rockingham Memorial Hospital Hahn Cancer Center, Harrisonburg, Virginia
  - Lynchburg Hematology-Oncology Clinic, Lynchburg, Virginia
  - Southwest VA Regional Cancer Center, Norton, Virginia
  - Auburn Regional Medical Center, Auburn, Washington
  - PeaceHealth Saint Joseph Medical Center, Bellingham, Washington
  - Harrison HealthPartners Hematology and Oncology-Bremerton, Bremerton, Washington
  - Providence Centralia Hospital, Centralia, Washington
  - Saint Francis Hospital, Federal Way, Washington
  - Columbia Basin Hematology and Oncology PLLC, Kennewick, Washington
  - Providence - Saint Peter Hospital, Olympia, Washington
  - Good Samaritan Community Hospital, Puyallup, Washington
  - Minor and James Medical PLLC, Seattle, Washington
  - Group Health Cooperative-Seattle, Seattle, Washington
  - Swedish Medical Center-First Hill, Seattle, Washington
  - The Polyclinic, Seattle, Washington
  - University of Washington Medical Center, Seattle, Washington
  - Cancer Care Northwest - Spokane South, Spokane, Washington
  - Rockwood Clinic, Spokane, Washington
  - Allenmore Hospital, Tacoma, Washington
  - Northwest CCOP, Tacoma, Washington
  - Saint Joseph Medical Center, Tacoma, Washington
  - Multicare Health System, Tacoma, Washington
  - Madigan Army Medical Center, Tacoma, Washington
  - Saint Clare Hospital, Tacoma, Washington
  - PeaceHealth Southwest Medical Center, Vancouver, Washington
  - Compass Oncology Vancouver, Vancouver, Washington
  - Camden-Clark Memorial Hospital, Parkersburg, West Virginia
  - Marshfield Clinic Cancer Center at Sacred Heart, Eau Claire, Wisconsin
  - Sacred Heart Hospital, Eau Claire, Wisconsin
  - Aurora Cancer Care-Southern Lakes, Elkhorn, Wisconsin
  - Agnesian Cancer Center, Fond du Lac, Wisconsin
  - Aurora Cancer Care-Glendale, Glendale, Wisconsin
  - Green Bay Oncology at Saint Vincent Hospital, Green Bay, Wisconsin
  - Saint Vincent Hospital, Green Bay, Wisconsin
  - Green Bay Oncology Limited at Saint Mary's Hospital, Green Bay, Wisconsin
  - Saint Mary's Hospital, Green Bay, Wisconsin
  - Mercy Health System, Janesville, Wisconsin
  - Mayo Clinic Health System-Franciscan Healthcare, La Crosse, Wisconsin
  - Bay Area Medical Center, Marinette, Wisconsin
  - Marshfield Clinic, Marshfield, Wisconsin
  - Saint Joseph's Hospital, Marshfield, Wisconsin
  - Medical Consultants Limited, Milwaukee, Wisconsin
  - Marshfield Clinic-Minocqua Center, Minocqua, Wisconsin
  - Green Bay Oncology - Oconto Falls, Oconto Falls, Wisconsin
  - Marshfield Clinic at James Beck Cancer Center, Rhinelander, Wisconsin
  - Marshfield Clinic-Rice Lake Center, Rice Lake, Wisconsin
  - Vince Lombardi Cancer Clinic-Sheboygan, Sheboygan, Wisconsin
  - Saint Michael's Hospital, Stevens Point, Wisconsin
  - Green Bay Oncology - Sturgeon Bay, Sturgeon Bay, Wisconsin
  - Marshfield Clinic-Wausau Center, Wausau, Wisconsin
  - Marshfield Clinic - Weston Center, Weston, Wisconsin
  - Marshfield Clinic - Wisconsin Rapids Center, Wisconsin Rapids, Wisconsin
  - Welch Cancer Center, Sheridan, Wyoming
- Canada (14):
  - Cross Cancer Institute, Edmonton, Alberta
  - Atlantic Health Sciences Corporation-Saint John Regional Hospital, Saint John, New Brunswick
  - Grand River Regional Cancer Centre at Grand River Hospital, Kitchener, Ontario
  - London Regional Cancer Program, London, Ontario
  - Credit Valley Hospital, Mississauga, Ontario
  - Lakeridge Health Oshawa, Oshawa, Ontario
  - Ottawa Health Research Institute-General Division, Ottawa, Ontario
  - Thunder Bay Regional Health Science Centre, Thunder Bay, Ontario
  - Saint Michael's Hospital, Toronto, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario
  - CSSS Champlain-Charles Le Moyne, Greenfield Park, Quebec
  - CHUQ - Pavilion Hotel-Dieu de Quebec, Québec, Quebec
  - Allan Blair Cancer Centre, Regina, Saskatchewan
  - Saskatoon Cancer Centre, Saskatoon, Saskatchewan
- Instituto Nacional de Enfermedades Neoplasicas, Lima, Peru
- Puerto Rico (2):
  - I Gonzales Martinez-Oncologic Hospital, San Juan
  - San Juan City Hospital, San Juan

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data may be made available upon request as per the ECOG-ACRIN Data Sharing Policy.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was activated on February 17, 2006 and accrued its first patient on May 11, 2006. Due to slow accrual, it was terminated on April 29, 2009 before reaching its accrual goal with final accrual of 355 patients.
Groups:
- Arm I (Oxaliplatin, Fluorouracil, Leucovorin): Patients receive oxaliplatin IV over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV on day 1 followed by fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment repeats every 2 weeks for up to 12 courses.
  oxaliplatin: Given IV
  fluorouracil: Given IV
  leucovorin calcium: Given IV
- Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab): Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive oxaliplatin, leucovorin calcium, and fluorouracil as in arm I.
  oxaliplatin: Given IV
  fluorouracil: Given IV
  leucovorin calcium: Given IV
  bevacizumab: Given IV
Period: Overall Study
Arm/Group | Arm I (Oxaliplatin, Fluorouracil, Leucovorin) | Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab)
Started | 176 | 179
Eligible | 171 | 177
Treated | 173 | 174
Completed | 126 | 106
Not Completed | 50 | 73
Not completed — Disease progression | 0 | 1
Not completed — Adverse Event | 26 | 36
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 11 | 20
Not completed — Alternative therapy | 2 | 0
Not completed — Other complicating disease | 0 | 1
Not completed — Not start protocol therapy | 3 | 5
Not completed — Other | 8 | 9

BASELINE CHARACTERISTICS:
Population: All randomized patients (intent-to-treat population)
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Oxaliplatin, Fluorouracil, Leucovorin) | Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab) | Total
Number analyzed (Participants) | 176 | 179 | 355
Age, Continuous [Median (Full Range); unit: Years] | 54 [22 to 80] | 53 [21 to 74] | 53 [21 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 62 | 67 | 129
  Male | 114 | 112 | 226

OUTCOME MEASURES:

1. Primary Outcome: 5-year Overall Survival Rate
Description: Overall survival (OS) was defined as time from randomization to date of death from any cause. Patients who were still alive were censored at last date of known alive. Kaplan-Meier method was used to estimate the 5-year OS rate.
Time Frame: Follow-up assessments performed every 3 months for patients < 2 years from randomization, every 6 months for patients 2-5 years from randomization, and every 12 months for patients 5-10 years from randomization
Population: All randomized patients (intent-to-treat population)
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Oxaliplatin, Fluorouracil, Leucovorin) | Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab)
Number analyzed (Participants) | 176 | 179
proportion of participants | 0.883 [0.523 to 0.924] | 0.837 [0.771 to 0.886]
Statistical Analysis 1: Comparison: Arm I (Oxaliplatin, Fluorouracil, Leucovorin) vs Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab); Test type: Superiority or Other; p = 0.876, Log Rank — Stratified log rank test. The above P value was for one-sided test

2. Secondary Outcome: 5-year Disease-free Survival Rate
Description: Disease-free survival (DFS) was defined as time from randomization to recurrence, second invasive primary cancer or death, whichever occurred first. Patients who were still alive and had no DFS events were censored at the last disease assessment date known to be free of DFS events. Kaplan-Meier method was used to estimate 5-year DFS rate.
Time Frame: as for outcome 1
Population: All randomized patients (intent-to-treat population)
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Arm I (Oxaliplatin, Fluorouracil, Leucovorin) | Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab)
Number analyzed (Participants) | 176 | 179
proportion of participants | 0.712 [0.634 to 0.776] | 0.765 [0.692 to 0.823]
Statistical Analysis 1: Comparison: Arm I (Oxaliplatin, Fluorouracil, Leucovorin) vs Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab); Test type: Superiority or Other; p = 0.299, Log Rank — two-sided stratified log rank test p value

3. Secondary Outcome: Patterns of Failure
Description: Failure included recurrence, second primary cancer and death without recurrence.
Time Frame: as for outcome 1
Population: all randomized patients
Measure: Number; unit: participants
Arm/Group | Arm I (Oxaliplatin, Fluorouracil, Leucovorin) | Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab)
Number analyzed (Participants) | 176 | 179
participants
  Local/regional recurrence | 6 | 5
  Distant recurrence | 24 | 20
  Mutiple recurrence | 5 | 8
  Unknown site | 1 | 1
  Death without recurrence | 5 | 6
  Second invasive primary cancer | 12 | 4
  DFS event | 52 | 41

4. Secondary Outcome: Proportion of Patients Who Completed 12 Cycles of Treatment
Description: In the study, treatment was repeated every 2 weeks for a total of 12 cycles on both arms. The total number of cycles of treatment patient received until going off treatment due to any reason was recorded. It was a measure of the tolerance of the therapy.
Time Frame: assessed at the end of treatment
Population: Patients who received at least one cycle of protocol treatment
Measure: Number; unit: proportion of participants
Arm/Group | Arm I (Oxaliplatin, Fluorouracil, Leucovorin) | Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab)
Number analyzed (Participants) | 173 | 174
proportion of participants | 0.722 | 0.615

5. Other Pre Specified Outcome: Change in Rectal Function Between Baseline and 12 Months
Description: Change in rectal function between baseline and 12 months was measuring the long-term rectal function among the patients. Rectal function was measured using the Bowel Function Questionnaire at baseline and 12 months after randomization. The total score of the questionnaire was calculated as the number of problems with bowel function (score range 0-11). Change in rectal function between baseline and 12 months= total score at 12 months - total score at baseline. A negative value indicated improved rectal function. This change in score was calculated for each individual patient who had the data.
Time Frame: assessed at baseline and 12 months after randomization
Population: Patients with data about their rectal function measured using the Bowel Function Questionnaire at both baseline and 12 months after randomization. Due to the early termination of the trial, the sample size was quite small for the endpoint. Consequently, it was considered as an exploratory endpoint.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm I (Oxaliplatin, Fluorouracil, Leucovorin) | Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab)
Number analyzed (Participants) | 12 | 11
scores on a scale | -1.17 (3.19) | 1.18 (3.09)

6. Other Pre Specified Outcome: Change in Oxaliplatin-related Neurotoxicity Between Baseline and 12 Months
Description: Change in oxaliplatin-related neurotoxicity between baseline and 12 months was measuring the long-term symptom of oxaliplatin-related neurotoxicity among the patients. Oxaliplatin-related neurotoxicity was measured using the FACT/GOG-Ntx subscale at baseline and 12 months after randomization. The range of the total score of the scale was between 0 and 44, and lower values indicate higher neurotoxicity. Change in oxaliplatin-related neurotoxicity between baseline and 12 months= total score at 12 months - total score at baseline. A negative value indicated worsened symptom. This change in score was calculated for each individual patient who had the data.
Time Frame: assessed at baseline and 12 months after randomization
Population: Patients with data about their oxaliplatin-related neurotoxicity measured using FACT/GOG Ntx subscale at both baseline and 12 months after randomization. Due to the early termination of the trial, the sample size was quite small for the endpoint. Consequently, it was considered as an exploratory endpoint.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Arm I (Oxaliplatin, Fluorouracil, Leucovorin) | Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab)
Number analyzed (Participants) | 53 | 62
scores on a scale | -8.6 (8.1) | -9.5 (7.9)

ADVERSE EVENTS:
Time Frame: Assessed every cycle (1 cycle=2 weeks) while on treatment and for 30 days after the end of treatment
Description: Long-term follow up form was used to collect any severe (grade>=3) long term toxicity experienced after discontinuing protocol therapy and prior to diagnosis of progression/relapse if the toxicity has not been previously reported yet. It was assessed every 3 months <2 year, every 6 months 2-5 years, and annually 5-10 years after study activation.
Groups:
- Arm I (Oxaliplatin, Fluorouracil, Leucovorin): Patients receive oxaliplatin intravenously (IV) over 2 hours, leucovorin calcium IV over 2 hours, and fluorouracil IV on day 1 followed by fluorouracil IV continuously over 46 hours on days 1 and 2. Treatment repeats every 2 weeks for up to 12 courses* in the absence of disease progression or unacceptable toxicity.
- Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab): Patients receive bevacizumab IV over 30-90 minutes on day 1. Patients also receive oxaliplatin, leucovorin calcium, and fluorouracil as in arm I
Arm/Group | Arm I (Oxaliplatin, Fluorouracil, Leucovorin) | Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab)
Serious Adverse Events (participants affected / at risk) | 119/173 | 123/174
Other Adverse Events (participants affected / at risk) | 154/173 | 155/174
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Oxaliplatin, Fluorouracil, Leucovorin) (N=173) | Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab) (N=174)
Allergic reaction (Immune system disorders) | 2 | 4
Anemia (Blood and lymphatic system disorders) | 2 | 2
Leukocytes decreased (Investigations) | 49 | 37
Lymphopenia (Investigations) | 16 | 9
Neutrophils decreased (Investigations) | 63 | 51
Platelets decreased (Investigations) | 12 | 1
Cardiac-ischemia (Cardiac disorders) | 1 | 2
Hypertension (Vascular disorders) | 0 | 11
Cardiomyopathy, restrictive (Cardiac disorders) | 0 | 1
Fatigue (General disorders) | 12 | 19
Fever w/o neutropenia (General disorders) | 2 | 0
Weight gain (Investigations) | 1 | 0
Weight loss (Investigations) | 1 | 0
INR increased (Investigations) | 0 | 1
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 0 | 5
Wound - non-infectious (Injury, poisoning and procedural complications) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 4 | 5
Dehydration (Metabolism and nutrition disorders) | 7 | 8
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 16 | 20
Dysphagia (Gastrointestinal disorders) | 0 | 2
Enteritis (Gastrointestinal disorders) | 1 | 0
Fistula, Colon/cecum/appendix (Gastrointestinal disorders) | 0 | 1
Fistula, Rectum (Gastrointestinal disorders) | 0 | 2
Dyspepsia (Gastrointestinal disorders) | 0 | 1
Ileus (Gastrointestinal disorders) | 1 | 1
Leak, incl. anastomotic, Leak NOS (Injury, poisoning and procedural complications) | 0 | 1
Leak, incl. anastomotic, rectum (Injury, poisoning and procedural complications) | 0 | 1
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 2 | 2
Muco/stomatitis (symptom) pharynx (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 6 | 6
Obstruction, small bowel NOS (Gastrointestinal disorders) | 1 | 1
Proctitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 7 | 1
GI-other (Gastrointestinal disorders) | 0 | 2
Lower GI, hemorrhage NOS (Gastrointestinal disorders) | 1 | 3
Rectum, hemorrhage (Gastrointestinal disorders) | 2 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 2 | 4
Infection w/ gr3-4 neut, colon (Infections and infestations) | 1 | 1
Infection w/ gr3-4 neut, sinus (Infections and infestations) | 0 | 1
Infection w/ gr3-4 neut, skin (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, colon (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, joint (Infections and infestations) | 1 | 0
Infection Gr0-2 neut, pelvis NOS (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, soft tissue (Infections and infestations) | 0 | 1
Infection Gr0-2 neut, urinary tract (Infections and infestations) | 0 | 3
Infection w/ unk ANC bladder (Infections and infestations) | 1 | 0
Infection w/ unk ANC catheter related (Infections and infestations) | 0 | 1
Infection-other (Infections and infestations) | 0 | 2
Alanine aminotransferase increased (Investigations) | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 2
Hypocalcemia (Metabolism and nutrition disorders) | 1 | 1
Creatinine increased (Investigations) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 3 | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 4 | 3
Proteinuria (Renal and urinary disorders) | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 4
Fracture (Injury, poisoning and procedural complications) | 1 | 0
Osteonecrosis (avascular necrosis) (Musculoskeletal and connective tissue disorders) | 0 | 1
Ataxia (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 1
Laryngeal nerve dysfunction (Nervous system disorders) | 1 | 0
Leukoencephalopathy (Nervous system disorders) | 0 | 1
Depression (Psychiatric disorders) | 0 | 1
Neuropathy-motor (Nervous system disorders) | 1 | 1
Neuropathy-sensory (Nervous system disorders) | 26 | 31
Syncope (Nervous system disorders) | 2 | 1
Neurologic-other (Nervous system disorders) | 0 | 1
Tearing (Eye disorders) | 0 | 1
Ocular-other (Eye disorders) | 0 | 1
Abdomen, pain (Gastrointestinal disorders) | 1 | 4
Back, pain (Musculoskeletal and connective tissue disorders) | 1 | 1
Bone, pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Cardiac/heart, pain (Cardiac disorders) | 0 | 1
Chest/thoracic pain NOS (General disorders) | 1 | 2
Extremity-limb, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Gallbladder, pain (Hepatobiliary disorders) | 1 | 0
Head/headache (Nervous system disorders) | 1 | 1
Joint, pain (Musculoskeletal and connective tissue disorders) | 0 | 4
Neck, pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Rectum, pain (Gastrointestinal disorders) | 1 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 8
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Prolong intubation post pulm resection (Injury, poisoning and procedural complications) | 0 | 1
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary/Upper Respiratory-other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Incontinence urinary (Renal and urinary disorders) | 0 | 1
Obstruction-ureteral (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 2
Urinary frequency/urgency (Renal and urinary disorders) | 0 | 1
Urinary retention (Renal and urinary disorders) | 0 | 1
Secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Vascular access,Thrombosis/embolism (Injury, poisoning and procedural complications) | 1 | 2
Thrombosis/thrombus/embolism (Vascular disorders) | 4 | 9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Oxaliplatin, Fluorouracil, Leucovorin) (N=173) | Arm II (Oxaliplatin, Fluorouracil, Leucovorin, Bevacizumab) (N=174)
Allergic reaction (Immune system disorders) | 9 | 5
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 5 | 12
Anemia (Blood and lymphatic system disorders) | 106 | 103
Leukocytes decreased (Investigations) | 104 | 98
Lymphopenia (Investigations) | 19 | 22
Neutrophils decreased (Investigations) | 83 | 72
Platelets decreased (Investigations) | 92 | 48
Hypertension (Vascular disorders) | 8 | 29
Fatigue (General disorders) | 122 | 121
Insomnia (Psychiatric disorders) | 22 | 35
Rigors/chills (General disorders) | 8 | 9
Weight loss (Investigations) | 14 | 20
Dry skin (Skin and subcutaneous tissue disorders) | 13 | 9
Alopecia (Skin and subcutaneous tissue disorders) | 33 | 35
Hyperpigmentation (Skin and subcutaneous tissue disorders) | 2 | 9
Nail changes (Skin and subcutaneous tissue disorders) | 12 | 15
Rash/desquamation (Skin and subcutaneous tissue disorders) | 19 | 15
Hand-foot reaction (Skin and subcutaneous tissue disorders) | 20 | 26
Anorexia (Metabolism and nutrition disorders) | 47 | 45
Constipation (Gastrointestinal disorders) | 34 | 36
Dehydration (Metabolism and nutrition disorders) | 10 | 17
Diarrhea w/o prior colostomy (Gastrointestinal disorders) | 84 | 84
Dysphagia (Gastrointestinal disorders) | 11 | 13
Dyspepsia (Gastrointestinal disorders) | 19 | 12
Muco/stomatitis by exam, oral cavity (Gastrointestinal disorders) | 34 | 34
Muco/stomatitis (symptom) oral cavity (Gastrointestinal disorders) | 35 | 34
Nausea (Gastrointestinal disorders) | 98 | 100
Taste disturbance (Nervous system disorders) | 23 | 23
Vomiting (Gastrointestinal disorders) | 37 | 37
Nose, hemorrhage (Respiratory, thoracic and mediastinal disorders) | 13 | 35
Hypoalbuminemia (Metabolism and nutrition disorders) | 14 | 7
Alkaline phosphatase increased (Investigations) | 31 | 15
Alanine aminotransferase increased (Investigations) | 21 | 13
Aspartate aminotransferase increased (Investigations) | 37 | 20
Hyperglycemia (Metabolism and nutrition disorders) | 18 | 22
Hypokalemia (Metabolism and nutrition disorders) | 16 | 15
Proteinuria (Renal and urinary disorders) | 2 | 15
Hyponatremia (Metabolism and nutrition disorders) | 10 | 9
Neuropathy-sensory (Nervous system disorders) | 132 | 130
Tearing (Eye disorders) | 5 | 11
Abdomen, pain (Gastrointestinal disorders) | 19 | 20
Head/headache (Nervous system disorders) | 16 | 24
Joint, pain (Musculoskeletal and connective tissue disorders) | 15 | 26
Muscle, pain (Musculoskeletal and connective tissue disorders) | 9 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 10 | 11
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 16 | 26
Voice changes/dysarthria (Respiratory, thoracic and mediastinal disorders) | 7 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less